CLINICAL TRIAL: NCT02917317
Title: South China Prospective Cohort Study of Chronic Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Di Li, Ph.D, Sun Yat-sen University
Other Study IDs: ZXYZM-5
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Retention Blood ,Urine and Stool samples for biochemical tests, biomarkers, DNA and so on
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the risk factors and prediction biomarkers of chronic disease in adults aged 35-74 years.

DETAILED DESCRIPTION:
To investigate the risk factors and prediction biomarkers of chronic disease within adults aged 35-74 years in South China. Following up the incidence of major chronic disease including stroke, coronary heart disease, cancer, chronic obstructive pulmonary disease, diabetes and hypertension.

ELIGIBILITY:
Inclusion Criteria:

aged 35-74 years local residents or lived in local for 5 years more

Exclusion Criteria:

Malignancy Cognitive impairment that can not cooperate with investigation

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: aged 35-74 years local residents or lived in local for 5 years more,no gender perfomance
Sampling Method: Non-Probability Sample
Enrollment: 110000 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic disease | 4 years or more
  Incidence of chronic disease, including stroke, coronary heart disease, cancer, chronic obstructive pulmonary disease, diabetes and hypertension

SECONDARY OUTCOMES:
Outcome of chronic disease | 4 years or more
  Outcome and development of chronic disease
Death | 4 years or more
  Death caused by chronic disease
Incidence of other disease | 4 years or more
  Incidence of other disease,including hyperuricaemia,fatty liver disease and so on

CONTACTS AND LOCATIONS:
Overall Officials: Fan J Hua, Ph.D, Principal Investigator — School of Public Health,Nutrition and Food Hygiene,Sun Yat-sen University
Locations (1):
- Guangdong Provincial Key Laboratory of Food, Nutrition and Health, Department of Nutrition, School of Public Health, Sun Yat-Sen University (Northern Campus), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
do not share participants data